CLINICAL TRIAL: NCT05334667
Title: Comparison Between the Effect of Continuous Renal Replacement Therapy Versus Plasmapheresis on Mortality Rate in Aluminum Phosphide Poisoning; Randomized Controlled Study
Brief Title: CRRT Versus Plasmapheresis in Aluminum Phosphide Poisoning
Acronym: AlP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rabab Ahmed Samy Anwer, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aluminum phosphide poisoning
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Aluminium Phosphide Poisoning
Keywords: CRRT; Plasmapheresis

STUDY DESIGN:
Intervention Model Description: Comparison between using CRRT versus plasmapheresis in the management of aluminum phosphide poisoning and effect on mortality rate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) The trial will be planned that neither the doctors (investigator) nor the patients will be aware of the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Patients will receive routine management only.
  Interventions: Other: Routine management
- CRRT group (Active Comparator): Patients will receive CRRT and routine management.
  Interventions: Other: Routine management; Device: CRRT
- PPH group (Active Comparator): Patients will receive plasmapheresis and routine management.
  Interventions: Other: Routine management; Device: PPH

INTERVENTIONS:
Other: Routine management — Routine management
Device: CRRT — Prisma-flex (Gambro-Swedan) machine will be used to carry out both CRRT and PPH sessions. Each CRRT session continue for 72 hours, while PPH session continue for 4 hours.
  Arms: CRRT group
Device: PPH — Prisma-flex (Gambro-Swedan) machine will be used to carry out both CRRT and PPH sessions. Each CRRT session continue for 72 hours, while PPH session continue for 4 hours.
  Arms: PPH group

SUMMARY:
Aluminum phosphide (AlP) is a solid fumigant pesticide sold as tablets in use since the 1940s. It is considered to be an ideal pesticide because of its cheapness, efficiency, and easy availability in the market and is widely used as a grain preservative worldwide.The mortality in cases of aluminum phosphide poisoning varies between 60% and 90%, even in experienced and well-equipped hospitals. Patients mostly die due to cardiovascular collapse, refractory shock, severe acidemia, fulminant hepatic failure, and or adult respiratory distress syndrome.

Continuous renal replacement therapy (CRRT) is a slow and smooth continuous extracorporeal blood purification, which is designed to replicate depurative function of the kidney. It is usually implemented over 24 h to several days with an aim of gentle correction of fluid overload and removal of excess uremic toxins. Furthermore, many observational studies considered CRRT as the predominant form of RRT in the intensive care unit (ICU) for critically ill patients with AKI and/or multiorgan failure, along with acute brain injury or other causes of increased intracranial pressure or generalized brain edema. The effectiveness of CRRT is mainly due to its accurate volume control, steady acid-base and electrolyte correction, and achievement of hemodynamic stability in adults and pediatrics.

Plasmapheresis (PPH) can rapidly and effectively remove toxic substances and their potentially toxic metabolites from the blood compartment, especially those with high protein-binding. As the potential benefit of therapeutic plasma exchange is increasingly recognized, its use is becoming more widespread, and case reports have confirmed its value in the treatment of drug overdose. The application of plasmapheresis dramatically reversed the severe biochemical and clinical manifestations and was able to prevent serious co-occurrence.

DETAILED DESCRIPTION:
Seventy five (75) patients will be included in this study. They will be randomly allocated into three groups (25 patients | each)

1. Control Group (C Group): routine management.
2. CRRT Group: routine management + CRRT.
3. PPH Group: routine management + PPH.

Immediately after ICU admission:

All Patients will receive the routine management including:

* Care for airway, breathing and circulation.
* Intravenous fluids guided by central venous pressure measurement and vasopressors (Norepinephrine) IV infusion will be used to treat hypotension and refractory shock, intubation and mechanical ventilation in the following conditions: apnea, respiratory failure, hypoxia, inadequate ventilation, disruption of airway reflexes, disturbed conscious level (GCS <8).
* Phosphine excretion can be increased by maintaining adequate hydration and renal perfusion with intravenous fluids and low dose dopamine (4-6 μg/kg/min). Diuretics like furosemide can be given if systolic blood pressure is >90 mm Hg to enhance excretion as the main route of elimination of phosphine is renal.
* Correction of metabolic acidosis by intravenous sodium bicarbonate will also be considered in a dose of 50-100 mEq intravenously every 8 hour till the bicarbonate level rises to 18-20 mEq/L.
* Additionally, magnesium sulfate: 1g IV infusion every 1hr for the first 3 hrs, followed by 1-1.5 g every 6 hrs for 24 hrs was administered.
* Decontamination will be done by gastric lavage using normal saline mixed with sodium bicarbonate solution (2 ampoules sodium bicarbonate 25% added to each 500cc saline) in all Patients presented within 2 hrs of toxic ingestion. Then, a single (50 gm) dose of activated charcoal will be administered.

Then patients will receive either CRRT or PPH after confirmation of exposure to aluminum phosphide.

Peri-interventional evaluation: -

1. Time elapsed between exposure and start of management.
2. Standard vital signs (ABP, HR, Spo2, ETCO2). ECG and GCS are continuously monitored and documented.
3. Laboratory studies:

   1. Phosphine gas level in blood by gas chromatography: on admission and another sample after CRRT or PPH
   2. Tropnin levels immediately on admission and at the end of CRRT or PPH.
   3. ABG to assess acid base status and lactate levels. Basic sample on admission and serial samples every 2 hours after the start of CRRT or PPH for follow up, evaluation and assessment.

Prisma-flex (Gambro-Swedan) machine will be used to carry out both CRRT and PPH sessions. Each CRRT session continue for 72 hours, while PPH session continue for 4 hours. The need for another session will be evaluated by the SBP< 90 mmHg, lactate level >1mmol, acid base status; PH<7.35 and renal function; S. creatinine>2.

All participating patients will be observed until discharge from the hospital or death. Continuous monitoring and documentation of their vital signs, oxygen saturation, and conscious level will be done.

Parameters to be evaluated regularly

1. Laboratory studies

   * CBC, Coagulation profile (PT, PC, INR) if within normal, reassessment after 48 hours.
   * Liver function tests LFTs if within normal, reassessment after 48 hours.
   * Urea and creatinine will be assessed daily.
   * Troponin T and I if within normal, reassessment after 48 hours.
   * Blood glucose/ 4 hours for the first 48 hours then every 8 hours.
   * K, Mg, Ca will be assessed daily.
2. Standard monitoring: ABP, HR, Spo2, ETCO2 and ECG continuously.
3. 24 hours total urine output (UOP).

ELIGIBILITY:
Inclusion Criteria:

* Patients exposed to AlP poisoning of either sex.
* Critically ill with severe symptomatic acute AlP poisoning; SBP<90mmHg, PH<7.32 and HR<60 bpm.
* Age >18 year.

Exclusion Criteria:

* Refusal to consent participating research.
* Age <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 30 days
  Evaluation of the effect of CRRT versus PPH on mortality rate in acute AlP poisoning, (30 days mortality).

SECONDARY OUTCOMES:
ICU | 30 days
  ICU stay.
Morbidity | 30 days
  Thirty days morbidity: organ dysfunction secondary to poisoning (e.g. renal failure, pancreatitis, DM).
Sessions | 30 days
  Frequency of CRRT and PPH sessions that will be required for each patient.
Vasopressors | 30 days
  Requirement of vasopressors and or inotropic support.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan LT, Crowley RJ, Delliou D, Geyer R. Phosphine analysis in post mortem specimens following ingestion of aluminium phosphide. J Anal Toxicol. 1983 Jul-Aug;7(4):165-7. doi: 10.1093/jat/7.4.165. PMID 6314042
- [Background] Yan H, Chen H, Li Z, Shen M, Zhuo X, Wu H, Xiang P. Phosphine Analysis in Postmortem Specimens Following Inhalation of Phosphine: Fatal Aluminum Phosphide Poisoning in Children. J Anal Toxicol. 2018 Jun 1;42(5):330-336. doi: 10.1093/jat/bky005. PMID 29378027
- [Background] Navabi SM, Navabi J, Aghaei A, Shaahmadi Z, Heydari R. Mortality from aluminum phosphide poisoning in Kermanshah Province, Iran: characteristics and predictive factors. Epidemiol Health. 2018 May 27;40:e2018022. doi: 10.4178/epih.e2018022. eCollection 2018. PMID 29807406
- [Background] Bellomo R, Ronco C. Nomenclature for continuous renal replacement therapies. Critical Care Nephrology: Springer; 1998. p. 1169-76.
- [Background] Ronco C, Ricci Z. Renal replacement therapies: physiological review. Intensive Care Med. 2008 Dec;34(12):2139-46. doi: 10.1007/s00134-008-1258-6. Epub 2008 Sep 13. PMID 18791697
- [Background] Macedo E, Mehta RL. Continuous Dialysis Therapies: Core Curriculum 2016. Am J Kidney Dis. 2016 Oct;68(4):645-657. doi: 10.1053/j.ajkd.2016.03.427. Epub 2016 May 28. No abstract available. PMID 27241853
- [Background] Schutt RC, Ronco C, Rosner MH. The role of therapeutic plasma exchange in poisonings and intoxications. Semin Dial. 2012 Mar-Apr;25(2):201-6. doi: 10.1111/j.1525-139X.2011.01033.x. Epub 2012 Feb 22. PMID 22353434